CLINICAL TRIAL: NCT06679972
Title: Intrahepatic Cholestasis of Pregnancy and the Respiratory Challenges of Bile Acids Pneumonia in Neonates (The CHOLE-RESP Trial)
Brief Title: Impact of Intrahepatic Cholestasis of Pregnancy on Neonatal Respiratory Outcomes
Acronym: CHOLE-RESP
Status: Enrolling by invitation | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Niculae Lucia-Elena, Doctoral Student, Medical Resident Neonatologist, Carol Davila University of Medicine and Pharmacy
Other Study IDs: 34/15.10.2024
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Intrahepatic Cholestasis of Pregnancy; Respiratory Distress Syndrome, Newborn
Keywords: bile-acid pneumonia; cholestasis of pregnancy; intrahepatic cholestasis; RDS; respiratory distress syndrome
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Respiratory Distress Syndrome, Newborn; Cholestasis, Intrahepatic; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — Serum extracted after centrifugation, frozen at minus 50 degrees Celsius
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cholestasis Group: This group will include all neonates born to mothers with intrahepatic cholestasis of pregnancy.
- Control Group: This group will include controls, defined as neonates born to mothers with no liver diseases.

SUMMARY:
Intrahepatic cholestasis of pregnancy is a liver condition in late pregnancy, causing itching and high bile acid levels that return to normal after birth. Babies born to mothers with this condition may have a higher risk of breathing issues. Researchers suspect bile acids might lead to a specific type of lung problem in newborns, but more studies are needed to confirm this.

DETAILED DESCRIPTION:
Intrahepatic cholestasis of pregnancy is a hepatic complication that predominantly arises during the second or third trimester. It is characterized by serum bile acid levels above 10 micromol/L and persistent pruritus, which resolves after delivery. To date, it has been observed that respiratory distress syndrome occurs more frequently in neonates born to mothers with cholestasis of pregnancy, and a potential new entity, 'acute bile acid-induced pneumonia,' has been proposed, though statistical confirmation is lacking. Therefore, the investigators deem it imperative to conduct a study in the neonatal population to establish a definitive conclusion regarding neonatal pulmonary impairment secondary to maternal bile acid accumulation.

ELIGIBILITY:
CASE

Inclusion Criteria:

* mother with recent diagnosis of intrahepatic cholestasis of pregnancy (serum bile acids over 10 micromol/l in the last 7 days before birth), with informed consent given a few hours before giving birth
* ursodeoxycholic acid, independent of dosage or initiation of treatment
* neonates born in Clinical Hospital of Obstetrics and Gynecology "Prof.Dr. Panait Sirbu"

Exclusion Criteria:

* no informed consent
* serum bile acids under 10 micromol/l in the last 7 days before birth
* newborns transferred from other neonatal units

CONTROL

Inclusion Criteria:

* mother with no history of hepatic disease during or before the current pregnancy, with informed consent given a few hours before giving birth
* neonates born in Clinical Hospital of Obstetrics and Gynecology "Prof.Dr. Panait Sirbu", of similar gestational age/weight/sex at birth to corresponding neonates in the cholestasis group

Exclusion Criteria:

* ursodeoxycholic acid, independent of dosage or initiation of treatment (suspected hepatic disease/elevated transaminases)
* newborns transferred from other neonatal units, with different gestational age/weight/sex than cases

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include selected neonates born at term or preterm age, in a third degree neonatal unit in Bucharest, Romania (Clinical Hospital of Obstetrics and Gynecology "Prof.Dr. Panait Sirbu"). For the cholestasis group, the study population is represented by neonates born to mothers with intrahepatic cholestasis diagnosed during pregnancy. The control group will include neonates of similar gestational age/weight/sex at birth born to mothers with no hepatic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of epithelial injury | In the first 24 hours, at 2-3 days and at 7 days of life
  This trial wishes to evaluate if neonates born to mothers with intrahepatic cholestasis of pregnancy are prone to develop a more extensive epithelial injury compared to those of similar gestational age/birthweight/sex born to mothers with no liver disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital of Obstetrics and Gynecology "Prof. Dr. Panait Sârbu", Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No